CLINICAL TRIAL: NCT03258892
Title: Sarcoma Treatment Guide Pilot Study
Brief Title: Sarcoma Treatment Guide in Improving Self-Monitoring in Patients With Sarcoma Receiving Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, James Chen, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-16301; NCI-2017-01277 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2017-08-17; First posted 2017-08-23 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (STG pre-chemotherapy) (Experimental): Patients receive the STG before completing 4 courses of standard of care chemotherapy.
  Interventions: Other: Educational Intervention; Other: Quality-of-Life Assessment; Other: Survey Administration
- Arm B (STG post-chemotherapy initiation) (Experimental): Patients complete 2 courses of standard of care chemotherapy and then receive the STG before completing 2 additional courses of standard of care chemotherapy.
  Interventions: Other: Educational Intervention; Other: Quality-of-Life Assessment; Other: Survey Administration

INTERVENTIONS:
Other: Educational Intervention — Receive STG
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Survey Administration — Ancillary studies

SUMMARY:
This randomized pilot clinical trial studies how well the Sarcoma Treatment Guide works in improving self-monitoring in patients with sarcoma who are receiving chemotherapy. The Sarcoma Treatment Guide may help patients with sarcoma to be better informed, become more engaged with care, encourage communication, and to better manage side effects associated with chemotherapy treatments in order to improve quality of life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate whether symptom management and communication are improved in patients who are chemotherapy naive who receive a Sarcoma Treatment Guide as compared to those that have not.

SECONDARY OBJECTIVES:

I. To explore whether patients who have previously undergone chemotherapy benefit from a Sarcoma Treatment Guide (STG) in regard to symptom management and have improved communication between patient and providers.

II. To assess patient satisfaction with using the STG at the end of the trial.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive the STG before completing 4 courses of standard of care chemotherapy.

ARM B: Patients complete 2 courses of standard of care chemotherapy and then receive the STG before completing 2 additional courses of standard of care chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Be able to read, write, and understand English
* Sarcoma clinic patient
* About to begin either oral or cytotoxic chemotherapy

Exclusion Criteria:

* Received previous chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Symptom management and communication improvement in chemotherapy naive patients as measured by participant survey and tracking telephone calls | Up to 1 year
  Will keep notes of qualitative feedback provided by participants regarding the Sarcoma Treatment Guide (STG) obtained from the survey. Notes will be reviewed to identify common themes that will be considered when making revisions to the STG to be used by chemotherapy patients in the Sarcoma Clinic. Telephone calls will be calculated for each participant associated with symptoms such as nausea, vomiting, diarrhea, constipation, and pain. The calls will be logged to track quantity, reason and outcome of all participants. Symptoms ratings self-reported by patients will be tracked using the Numeri

SECONDARY OUTCOMES:
Patient satisfaction with Sarcoma Treatment Guide (STG) as measured by participant survey and tracking telephone calls | Up to 1 year
  Will keep notes of qualitative feedback provided by participants regarding the STG obtained from the survey. Notes will be reviewed to identify common themes that will be considered when making revisions to the STG to be used by chemotherapy patients in the Sarcoma Clinic. Telephone calls will be calculated for each participant associated with symptoms such as nausea, vomiting, diarrhea, constipation, and pain. The calls will be logged to track quantity, reason and outcome of all participants. Symptoms ratings self-reported by patients will be tracked using the NRS. Secondary analysis will inc
Sarcoma Treatment Guide (STG) benefit in patients who have undergone chemotherapy as measured by participant survey and tracking telephone calls | Up to 1 year
  Will keep notes of qualitative feedback provided by participants regarding the STG obtained from the survey. Notes will be reviewed to identify common themes that will be considered when making revisions to the STG to be used by chemotherapy patients in the Sarcoma Clinic. Telephone calls will be calculated for each participant associated with symptoms such as nausea, vomiting, diarrhea, constipation, and pain. The calls will be logged to track quantity, reason and outcome of all participants. Symptoms ratings self-reported by patients will be tracked using the NRS (Numeric Ratings Scale). Secondary analysis will inc

CONTACTS AND LOCATIONS:
Overall Officials: James Chen, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Speece NJ, Xu M, Tinoco G, Liebner DA, Chen JL. Randomized Prospective Trial Exploring the Impact of Structured Journaling in Patients With Sarcoma on the Management of Treatment-Related Adverse Events. JCO Oncol Pract. 2022 Feb;18(2):e250-e260. doi: 10.1200/OP.21.00309. Epub 2021 Sep 24. PMID 34559571
- See also: The Jamesline — http://cancer.osu.edu